CLINICAL TRIAL: NCT05775276
Title: Incidence Of Mesh Infection After Hernioplasty In Obstructed and Strangulated Hernia Using Proline Mesh and Sutures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Abdelnaeem, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Incidence Of Mesh Infection
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Incidence of Mesh Infection In Hernioplasty
MeSH Terms: interventions — Herniorrhaphy

STUDY DESIGN:
Intervention Model Description: All adult patients aging above 21 years old, who presented with obstructed or strangulated hernia with viable bowel loops by clinical examination or detected by preoperative ultrasound or computed tomography CT imaging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incidence Of Mesh Infection After proline mesh Hernioplasty (Experimental): Cases presented with strangulated or obstructed hernia
  Interventions: Procedure: Proline mesh in hernioplasty

INTERVENTIONS:
Procedure: Proline mesh in hernioplasty — Hernioplasty using proline mesh then follow up for incidence of infection

SUMMARY:
The primary aim of this study is to detect incidence of mesh infection in cases presented with obstructed or strandulated hernia.A prospective controlled study will be carried out after obtaining written informed consent from all patients and approval of the ethics committee of the faculty of medicine, Assuit University.

DETAILED DESCRIPTION:
There is controversy regarding the use of prolene mesh in cases of obstructed and strangulated hernia. The main aim and objective of this prospective study is to evaluate the outcomes and incidence of mesh infection in hernioplasty in emergency situations like obstructed and strangulated hernia .Hernioplasty is the most common surgery for hernia repair with Propylene mesh,but the use of synthetic prosthesis is associated with increase risk of developing a prosthetic infection that may manifest after time as subtle symptoms in the form of fever, myalgia, erythema of overlying skin and in some cases as chronic discharging sinus(1). clinicians have been challenged in the past few years by an increasing variety of novel non-infectious and infectious complications following the widespread use of meshes after open repair of hernias this incidence is influenced by underlying co-morbidities, the type of mesh, the surgical technique and the strategy used to prevent infections. An approach that combines medical and surgical management is necessary for cases of mesh infection.(2)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aging above 21 years old, who presented with obstructed or strangulated hernia with viable bowel loops by clinical examination or detected by preoperative ultrasound or computed tomography CT imaging.

Exclusion Criteria:

* Uncomplicated hernia.
* patients who will underwent rescection and anastmosis
* patient cannot withstand anethesia.
* Decompensated liver patients.
* Pregnancy.
* Immunosuppressed patients e.g.: under chemotherapy or steroids.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence Of Mesh Infection After Hernioplasty In Complicated Hernia Using Proline Mesh and Sutures | Baseline
  To evaluate the incidence of mesh infection in Complicated hernia using prolene mesh and sutures,along postoperative hospital stay, routine follow up and time to return to activities of daily living.

REFERENCES:
- [Result] Chung L, Tse GH, O'Dwyer PJ. Outcome of patients with chronic mesh infection following abdominal wall hernia repair. Hernia. 2014 Oct;18(5):701-4. doi: 10.1007/s10029-014-1277-x. Epub 2014 Jul 20. PMID 25038894
- [Result] Sanchez VM, Abi-Haidar YE, Itani KM. Mesh infection in ventral incisional hernia repair: incidence, contributing factors, and treatment. Surg Infect (Larchmt). 2011 Jun;12(3):205-10. doi: 10.1089/sur.2011.033. Epub 2011 Jul 18. PMID 21767146